CLINICAL TRIAL: NCT01225952
Title: A Three Arm Prospective Clinical Evaluation of Three FDA-approved Intraocular Lenses Designed to Improve Distance, Intermediate and Near Vision Following Lens Extraction
Brief Title: Three Intraocular Lenses Designed to Improve Distance, Intermediate and Near Vision Following Lens Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 656
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-12

CONDITIONS: Cataract
Keywords: phacoemulsification; intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Crystalens AO (Experimental): Bausch & Lomb silicone multi-piece accommodating IOL is a modified plate haptic lens
  Interventions: Device: Crystalens AO
- ReSTOR 3.0 (Active Comparator): An aspheric multifocal IOL (Alcon Laboratories) combines the functions of an apodized diffractive region and a refractive region.
  Interventions: Device: ReSTOR 3.0
- AMO Tecnis Multifocal (Active Comparator): A foldable hydrophobic acrylic IOL,(Abbott Medical Optics), is an ultraviolet light-absorbing posterior chamber IOL
  Interventions: Device: AMO Tecnis Multifocal

INTERVENTIONS:
Device: Crystalens AO — Bausch & Lomb model silicone multi-piece accommodating IOL.
  Arms: Crystalens AO
Device: ReSTOR 3.0 — An aspheric multifocal IOL (Alcon Laboratories) combines the functions of an apodized diffractive region and a refractive region.
  Arms: ReSTOR 3.0
Device: AMO Tecnis Multifocal — The Tecnis Multifocal foldable hydrophobic acrylic IOL, Model ZMA00 (Abbott Medical Optics), is an ultraviolet light-absorbing posterior chamber IOL.
  Arms: AMO Tecnis Multifocal

SUMMARY:
The objective of this study is to compare the contrast sensitivity, high and low contrast visual acuity (VA), glare meter outcomes, and subject satisfaction with three different FDA-approved intraocular lenses (IOLs) designed to improve distance, intermediate, and near vision following lens extraction in adults at least 40 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing primary IOL implantation for the correction of aphakia following continuous curvilinear anterior capsulotomy and phacoemulsification cataract extraction.
* Subjects must require a spherical lens power from 10.00 diopters (D) to 33.00 D.
* Subjects must have the potential for corrected distance visual acuity (CDVA) of 20/32 or better in both eyes.
* Subjects must have stopped contact lens wear for at least two weeks for soft lens wearers or three weeks for gas permeable lens wearers prior to biometry and surgery.
* At the time of surgery, subjects must have an intact centered capsulorhexis, intact posterior capsule, and no zonular rupture.
* Subjects must have ≤ 1.25 D of preoperative corneal astigmatism in both eyes.

Exclusion Criteria:

* Subjects with diagnoses of degenerative visual disorders (eg, macular degeneration, or other retinal disorders) that cause potential acuity losses to a level of 20/32 or worse.
* Subjects with conditions with increased risk of zonular rupture, such as pseudoexfoliation syndrome.
* Subjects who have any active inflammation or edema (swelling) of the cornea, including but not limited to the following: keratitis, keratoconjunctivitis, and keratouveitis.
* Subjects with uncontrolled glaucoma.
* Subjects with previous retinal detachment.
* Subjects with visually significant diabetic retinopathy (proliferative or nonproliferative) which reduces potential acuity to 20/32 or worse.
* Subjects with rubella, bilateral congenital, traumatic, complicated or polar cataract.
* Subjects with marked microphthalmos or aniridia.
* Subjects who have had previous corneal surgery.
* Subjects with irregular corneal astigmatism.
* Subjects with amblyopia which reduces potential acuity to 20/32 or worse.
* Subjects with optic atrophy.
* Subjects with iris neovascularization.
* Subjects with clinically significant retinal pigment epithelium/macular changes which reduces potential acuity to 20/32 or worse.
* Subjects with chronic use of systemic steroids or immunosuppressive medications.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tes Ignacio, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Asian Eye Institute, Makati City, Philippines

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an evaluation of three United States Food and Drug Administration (FDA) approved IOLs. A total of 93 participants(186 eyes) were enrolled at one investigative site in the Philippines. First participant was enrolled 7/15/2010 and last participant exited the study 4/28/2011.
Pre-assignment Details: 186 participant eyes were enrolled in this study 154 participant eyes completed the study. Participants underwent bilateral phacoemulsification and IOL implantation. Participants were randomized to treatment groups prior to surgery.
Period: Overall Study
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Started | 31 | 31 | 31
Completed | 25 | 27 | 25
Not Completed | 6 | 4 | 6
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Study Eye Explanted | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 5
Not completed — Surgical complications | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal | Total
Number analyzed (Participants) | 31 | 31 | 31 | 93
Age, Customized [Number; unit: participants]
  < 40 years | 0 | 0 | 0 | 0
  40 - 49 years | 2 | 1 | 0 | 3
  50 - 59 years | 6 | 8 | 7 | 21
  60 - 69 years | 13 | 14 | 16 | 43
  70 - 79 years | 10 | 8 | 7 | 25
  >/= 80 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 22 | 70
  Male | 8 | 6 | 9 | 23
Region of Enrollment [Number; unit: participants]
  Philippines | 31 | 31 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare (1.5, 3 Cycles/Degree)
Description: A single eye (monocular) in dim light (mesopic) measuring contrast sensitivity; The participant is presented with a sine-wave grating target of a given spatial frequency (cycles/degree of visual angle) where the smaller the number of cycles/degree the wider apart the gradations (vertical lines of grayness). The participant's ability to detect changes in contrast is determined. Higher mean indicates improved contrast sensitivity.
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 26 | 27 | 25
Number analyzed (eyes) | 52 | 54 | 50
log contrast sensitivity units
  1.5 cycles/degree | 1.612 (0.229) | 1.582 (0.231) | 1.527 (0.248)
  3 cycles/degree | 1.658 (0.195) | 1.627 (0.224) | 1.629 (0.240)

2. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare(6 Cycles/Degree)
Description: as for outcome 1
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set, non-missing
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 26 | 25 | 24
Number analyzed (eyes) | 51 | 50 | 48
log contrast sensitivity units | 1.641 (0.210) | 1.611 (0.237) | 1.641 (0.286)

3. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(1.5, 3 Cycles/Degree)
Description: In two eye (Binocular) in dim light (mesopic) measuring contrast sensitivity; The participant is presented with a sine-wave grating target of a given spatial frequency (cycles/degree of visual angle) where the smaller the number of cycles/degree the wider apart the gradations (vertical lines of grayness). The participant's ability to detect changes in contrast is determined. Higher mean indicates improved contrast sensitivity.
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 26 | 27 | 25
log contrast sensitivity units
  1.5 cycles/degree | 1.770 (0.187) | 1.656 (0.238) | 1.605 (0.203)
  3 cycles/degree | 1.807 (0.199) | 1.679 (0.275) | 1.689 (0.189)

4. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(6 Cycles/Degree)
Description: In two eyes (binocular) in dim light (mesopic) measuring contrast sensitivity; The participant is presented with a sine-wave grating target of a given spatial frequency (cycles/degree of visual angle) where the smaller the number of cycles/degree the wider apart the gradations (vertical lines of grayness). The participant's ability to detect changes in contrast is determined. Higher mean indicates improved contrast sensitivity.
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 25 | 26 | 25
log contrast sensitivity units | 1.825 (0.216) | 1.591 (0.274) | 1.700 (0.284)

5. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare(12 Cycles/Degree)
Description: as for outcome 1
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set, non-missing
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 24 | 22 | 21
Number analyzed (eyes) | 48 | 43 | 42
log contrast sensitivity units | 1.325 (0.226) | 1.227 (0.198) | 1.324 (0.281)

6. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare(18 Cycles/Degree)
Description: as for outcome 1
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set, non-missing
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 17 | 13 | 15
Number analyzed (eyes) | 34 | 26 | 30
log contrast sensitivity units | 0.977 (0.266) | 0.985 (0.185) | 0.973 (0.342)

7. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare(1.5, 3 Cycles/Degree)
Description: as for outcome 1
Time Frame: Postoperative visit 4 (day 120-180)
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 25 | 27 | 25
Number analyzed (eyes) | 50 | 54 | 50
log contrast sensitivity units
  1.5 cycles/degree | 1.696 (0.213) | 1.621 (0.222) | 1.527 (0.190)
  3 cycles/degree | 1.678 (0.159) | 1.670 (0.236) | 1.630 (0.203)

8. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare(6 Cycles/Degree)
Description: as for outcome 1
Time Frame: Postoperative visit 4 (day 120-180)
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 24 | 26 | 24
Number analyzed (eyes) | 48 | 51 | 48
log contrast sensitivity units | 1.579 (0.239) | 1.499 (0.230) | 1.610 (0.228)

9. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare(12 Cycles/Degree)
Description: as for outcome 1
Time Frame: Postoperative visit 4 (day 120-180)
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 20 | 18 | 20
Number analyzed (eyes) | 39 | 35 | 40
log contrast sensitivity units | 1.280 (0.245) | 1.225 (0.253) | 1.230 (0.248)

10. Primary Outcome: Monocular Mesopic Contrast Sensitivity Without Glare(18 Cycles/Degree)
Description: as for outcome 1
Time Frame: Postoperative visit 4 (day 120-180)
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 13 | 10 | 9
Number analyzed (eyes) | 25 | 20 | 18
log contrast sensitivity units | 0.974 (0.303) | 0.980 (0.246) | 0.976 (0.207)

11. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(12 Cycles/Degree)
Description: as for outcome 4
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 25 | 21 | 22
log contrast sensitivity units | 1.425 (0.221) | 1.335 (0.218) | 1.361 (0.278)

12. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(18 Cycles/Degree)
Description: as for outcome 4
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 19 | 15 | 16
log contrast sensitivity units | 1.029 (0.250) | 1.001 (0.213) | 0.981 (0.362)

13. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(1.5, 3 Cycles/Degree)
Description: as for outcome 4
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 25 | 27 | 25
log contrast sensitivity units
  1.5 cycles/degree | 1.797 (0.183) | 1.751 (0.238) | 1.577 (0.206)
  3 cycles/degree | 1.851 (0.178) | 1.723 (0.239) | 1.702 (0.219)

14. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(6 Cycles/Degree)
Description: as for outcome 4
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 24 | 25 | 24
log contrast sensitivity units | 1.758 (0.280) | 1.640 (0.236) | 1.690 (0.263)

15. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(12 Cycles/Degree)
Description: as for outcome 4
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 21 | 18 | 22
log contrast sensitivity units | 1.371 (0.247) | 1.269 (0.257) | 1.310 (0.286)

16. Secondary Outcome: Binocular Mesopic Contrast Sensitivity Without Glare(18 Cycles/Degree)
Description: as for outcome 4
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 16 | 12 | 12
log contrast sensitivity units | 1.115 (0.299) | 0.995 (0.384) | 1.041 (0.330)

17. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(1.5 Cycles/Degree)
Description: In one eye (monocular) in dim light (mesopic) measuring contrast sensitivity; The participant is presented with a sine-wave grating target of a given spatial frequency (cycles/degree of visual angle) where the smaller the number of cycles/degree the wider apart the gradations (vertical lines of grayness). The participant's ability to detect changes in contrast is determined. Higher mean indicates improved contrast sensitivity.
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 26 | 25 | 25
Number analyzed (eyes) | 52 | 50 | 49
log contrast sensitivity units | 1.591 (0.215) | 1.519 (0.218) | 1.482 (0.268)

18. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare (3 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 26 | 25 | 24
Number analyzed (eyes) | 52 | 50 | 47
log contrast sensitivity units | 1.687 (0.229) | 1.581 (0.204) | 1.588 (0.264)

19. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(6 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 25 | 25 | 23
Number analyzed (eyes) | 50 | 49 | 45
log contrast sensitivity units | 1.674 (0.237) | 1.531 (0.238) | 1.626 (0.293)

20. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(12 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 23 | 18 | 17
Number analyzed (eyes) | 45 | 35 | 34
log contrast sensitivity units | 1.328 (0.224) | 1.230 (0.223) | 1.340 (0.268)

21. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(18 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 3 (day 30-60)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 14 | 12 | 13
Number analyzed (eyes) | 27 | 24 | 25
log contrast sensitivity units | 1.024 (0.196) | 0.945 (0.158) | 0.834 (0.283)

22. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(1.5 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 25 | 25 | 24
Number analyzed (eyes) | 50 | 50 | 48
log contrast sensitivity units | 1.550 (0.263) | 1.488 (0.226) | 1.449 (0.206)

23. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(3 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 25 | 25 | 25
Number analyzed (eyes) | 50 | 50 | 49
log contrast sensitivity units | 1.664 (0.258) | 1.572 (0.225) | 1.535 (0.220)

24. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(6 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 24 | 23 | 23
Number analyzed (eyes) | 48 | 46 | 45
log contrast sensitivity units | 1.578 (0.252) | 1.493 (0.267) | 1.519 (0.260)

25. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(12 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 20 | 15 | 16
Number analyzed (eyes) | 39 | 30 | 31
log contrast sensitivity units | 1.335 (0.298) | 1.246 (0.278) | 1.194 (0.237)

26. Secondary Outcome: Monocular Mesopic Contrast Sensitivity With Glare(18 Cycles/Degree)
Description: as for outcome 17
Time Frame: Postoperative visit 4 (day 120-180)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: log contrast sensitivity units
Units Other Than Participants: eyes
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Number analyzed (Participants) | 13 | 8 | 8
Number analyzed (eyes) | 25 | 16 | 16
log contrast sensitivity units | 0.919 (0.283) | 1.019 (0.367) | 0.935 (0.207)

ADVERSE EVENTS:
Time Frame: 120-180 days
Description: Adverse events measured by eye
Arm/Group | Crystalens AO | ReSTOR 3.0 | AMO Tecnis Multifocal
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 12/53 | 5/54 | 6/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystalens AO (N=53) | ReSTOR 3.0 (N=54) | AMO Tecnis Multifocal (N=51)
Increased Intraocular Pressure (Eye disorders) | 11 (11) | 5 (5) | 3 (3)
Cystoid Macular Edema (Eye disorders) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s)after the review by, and in consultation and agreement with the Sponsor.